CLINICAL TRIAL: NCT00249093
Title: Effects of Supplementary Oxygen on Dyspnoea and Exercise Tolerance in COPD Patients Given LTOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Collaborators: The norwegian association for heart and lung patients (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: G25-1
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oxygen

SUMMARY:
The aim of the study is to evaluate effects of supplementary oxygen during exercise on dyspnoea and exercise tolerance in COPD-patients given long-time oxygen treatment

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (male/female)given long-term oxygen treatment
* Able to perform two separate walking tests

Exclusion Criteria:

* Severe heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2005-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
dyspnea
exercise tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Morten S Ryg, dr philos, Principal Investigator — LHL Helse
Locations (1):
- Glittreklinikken, Hakadal, Hakadal, Norway